CLINICAL TRIAL: NCT04557475
Title: A Randomized Trial of Transplacental Aspirin Therapy for Early Onset Fetal Growth
Brief Title: Transplacental Aspirin Therapy for Early Onset Fetal Growth Restriction
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We are modifying this trial's protocol and will resubmit a new application at a later date.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00259253
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Fetal Growth Restriction; Fetal Growth Retardation; Intrauterine Growth Restriction; Intrauterine Growth Retardation
Keywords: Maternal Aspirin Therapy
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Two Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASA Group (Experimental): Receives standard of care and intervention.
  Interventions: Drug: Aspirin
- SOC Group (No Intervention): Receives standard of care (SOC), only

INTERVENTIONS:
Drug: Aspirin — Two tablets daily with dinner
  Other Names: acetylsalicylic acid (ASA)
  Arms: ASA Group

SUMMARY:
The purpose of this investigation is to evaluate the ability of maternal aspirin (ASA) therapy to prevent preterm birth for fetal indications prior to 32 weeks gestation in women with early onset Fetal Growth Restriction (FGR). Aspirin is a commonly used medication that blocks blood platelets from clumping. Aspirin crosses the placenta in a dose dependent mode. There is preliminary evidence in smaller studies that aspirin can block fetal platelet clumping and, therefore, slow down the progression of placental disease under specific circumstances. The optimal time for aspirin to work is when the fetus' placental dysfunction is still mild. The goal of this research study is to show if fetuses that receive aspirin through maternal intake at a dose shown to affect fetal platelet aggregation will be less likely to deliver before 32 weeks for fetal deterioration. The outcomes of patients that receive aspirin will be compared to women that receive standard FGR management but do not take any aspirin. The decision if a study participant receives aspirin or not will be randomly picked. Such a research study is called a randomized controlled trial.

DETAILED DESCRIPTION:
Early onset FGR requiring preterm delivery by 32 weeks gestation complicates 1-5% of pregnancies and is an important health problem. Over 60% of children have long-term health consequences after being delivered for early onset FGR. There is no prenatal treatment for fetal growth restriction. The current management of FGR consists of fetal surveillance to detect a decline in the baby's health and deliver when this can be safely done. In a large number of early onset FGR, premature delivery is required to prevent the fetus from becoming more compromised or even dying in the womb.

Placental dysfunction leading to early onset FGR is characterized by changes to the blood vessels of the placenta, leading to a decline in the amount of blood flow to the placenta. The arteries that run in the umbilical cord of the fetus (umbilical arteries) are important for nutrient exchange between the fetal and placental circulation. Many fetuses with early onset FGR have elevated resistance in the blood vessels entering the placenta. This results in decreased blood flow in the umbilical artery (UA). The blood flow in the umbilical artery is evaluated by a specialized ultrasound technique called Doppler ultrasound. Doppler ultrasound of the umbilical arteries examines the blood flow to see if there is evidence of abnormal blood flow into the placenta. When the amount of blood flow at the end of every pulse decreases, it is classified as elevated UA blood flow resistance. When the blood flow briefly pauses at the end of each pulse, this is called absent end-diastolic velocity (AEDV) or UA AEDV. When the blood flow reverses at the end of each pulse, this is called reversed end-diastolic velocity (UA REDV). In fetuses with elevated UA blood flow, the placenta can usually supply enough nutrients and oxygen for at least 9 weeks. After that time, delivery is typically required. The worsening of blood flow to UA AEDV, or even UA REDV, increases the risk for fetal deterioration and preterm birth within the next 2-6 weeks. Approximately, 80% of early onset FGR fetuses progress to UA AEDV, or even UA REDV, and then require delivery by 32 weeks. There is no treatment that can stop this progression which is of critical importance in determining how much time is left for the fetus before delivery will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years old
* Gestational age between 220/7 to 300/7 weeks
* Fetal abdominal circumference < 10th percentile
* Umbilical artery Doppler index elevation > 95th percentile
* Forward umbilical artery end-diastolic flow
* Able to understand purpose, risks/benefits, and voluntary nature of study participant

Exclusion Criteria:

* Multiple pregnancy
* Currently taking 81 mg aspirin
* Maternal contraindication to aspirin treatment including allergy
* Active vaginal bleeding
* Presence of any physical fetal anomaly
* Fetal viral infection if diagnosed by the appropriate diagnostic test
* Fetal chromosomal abnormalities if diagnosed by invasive fetal testing
* Need for imminent delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-11 (Estimated); Primary Completion 2023-06-11 (Estimated); Study Completion 2023-06-11 (Estimated)

PRIMARY OUTCOMES:
Number of fetuses delivered for non-reassuring fetal status prior to 32+0 week's gestation | From randomization until birth, up to 38 weeks gestation
  To determine the frequency of delivery prior to 32+0 weeks' gestation for abnormal fetal surveillance parameters.

SECONDARY OUTCOMES:
Change in UA Doppler index | Baseline and weekly, up to 38 weeks gestation
  UA Doppler index is assessed at enrollment (baseline) and weekly. Qualitative changes in UA Doppler index are measured as presence, absence or reversal of end-diastolic velocity.
Change in amniotic fluid index (AFI) | Baseline and weekly, up to 38 weeks gestation
  Amniotic fluid index, measured with amniotic fluid volume [in centimeters (cm)] will be assessed at enrollment (baseline) and weekly. Oligohydramnios is an AFI ≤ 5 cm or a maximum vertical pocket (MVP) pocket ≤ 2 cm.
Change in fetal heart rate decelerations | Baseline and weekly to bi-weekly, up to 38 weeks gestation
  Fetal heart rate decelerations [in milliseconds (ms)] is assessed at enrollment (baseline) and weekly to bi-weekly. Heart rate variability increases with gestational age. After 29 weeks gestation, 4.0 ms and 3.0 ms meet criteria for reduced or very low short-term variation (STV) respectively. Before 29 weeks gestation, an STV <3.5 ms is considered reduced and <2.6 ms as very low.
Change in biophysical profile score | Baseline and weekly to bi-weekly, up to 38 weeks gestation
  Biophysical profile score is assessed at enrollment (baseline) and weekly to bi-weekly. The biophysical profile (BPP) combines a nonstress test (NST) with an ultrasound to evaluate a baby's heart rate, breathing, movements, muscle tone and amniotic fluid level. Each gives a score between 0 and 2 and are added up for a total maximum score of 10. A score of 8 or 10 is considered normal, while a score below 8 usually requires further evaluation or delivery of the baby.
Gestational age at delivery | At time of birth, up to 38 weeks gestation
  Gestational age at delivery measured in weeks.
Birthweight percentile at delivery | At time of birth, up to 38 weeks gestation
  Birthweight percentile will be assessed at the time of delivery.
Placental size at delivery | At time of birth, up to 38 weeks gestation
  Placental size measured in grams at delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet A Baschat, Principal Investigator — Johns Hopkins University; Ashi R Daftary, MD, Principal Investigator — Allegheny Health Network

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khong TY, Mooney EE, Ariel I, Balmus NC, Boyd TK, Brundler MA, Derricott H, Evans MJ, Faye-Petersen OM, Gillan JE, Heazell AE, Heller DS, Jacques SM, Keating S, Kelehan P, Maes A, McKay EM, Morgan TK, Nikkels PG, Parks WT, Redline RW, Scheimberg I, Schoots MH, Sebire NJ, Timmer A, Turowski G, van der Voorn JP, van Lijnschoten I, Gordijn SJ. Sampling and Definitions of Placental Lesions: Amsterdam Placental Workshop Group Consensus Statement. Arch Pathol Lab Med. 2016 Jul;140(7):698-713. doi: 10.5858/arpa.2015-0225-CC. Epub 2016 May 25. PMID 27223167
- [Background] Kingdom JC, Burrell SJ, Kaufmann P. Pathology and clinical implications of abnormal umbilical artery Doppler waveforms. Ultrasound Obstet Gynecol. 1997 Apr;9(4):271-86. doi: 10.1046/j.1469-0705.1997.09040271.x. No abstract available. PMID 9168580
- [Background] Morrow RJ, Adamson SL, Bull SB, Ritchie JW. Effect of placental embolization on the umbilical arterial velocity waveform in fetal sheep. Am J Obstet Gynecol. 1989 Oct;161(4):1055-60. doi: 10.1016/0002-9378(89)90783-7. PMID 2679101
- [Background] Giles WB, Trudinger BJ, Baird PJ. Fetal umbilical artery flow velocity waveforms and placental resistance: pathological correlation. Br J Obstet Gynaecol. 1985 Jan;92(1):31-8. doi: 10.1111/j.1471-0528.1985.tb01045.x. PMID 3966988
- [Background] Jackson MR, Walsh AJ, Morrow RJ, Mullen JB, Lye SJ, Ritchie JW. Reduced placental villous tree elaboration in small-for-gestational-age pregnancies: relationship with umbilical artery Doppler waveforms. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):518-25. doi: 10.1016/0002-9378(95)90566-9. PMID 7856679
- [Background] Redline RW, Ravishankar S. Fetal vascular malperfusion, an update. APMIS. 2018 Jul;126(7):561-569. doi: 10.1111/apm.12849. PMID 30129125
- [Background] Wilcox GR, Trudinger BJ. Fetal platelet consumption: a feature of placental insufficiency. Obstet Gynecol. 1991 Apr;77(4):616-21. PMID 2002988
- [Background] Trudinger B, Song JZ, Wu ZH, Wang J. Placental insufficiency is characterized by platelet activation in the fetus. Obstet Gynecol. 2003 May;101(5 Pt 1):975-81. doi: 10.1016/s0029-7844(03)00173-x. PMID 12738160
- [Background] Ohshige A, Yoshimura T, Maeda T, Ito M, Okamura H. Increased platelet-activating factor-acetylhydrolase activity in the umbilical venous plasma of growth-restricted fetuses. Obstet Gynecol. 1999 Feb;93(2):180-3. doi: 10.1016/s0029-7844(98)00407-4. PMID 9932551
- [Background] Sciscione AC, Bessos H, Callan N, Blakemore K, Kickler T. Indicators of platelet turnover in thrombocytopenic infants. Br J Obstet Gynaecol. 1997 Jun;104(6):743-5. doi: 10.1111/j.1471-0528.1997.tb11990.x. PMID 9197883
- [Background] Baschat AA, Gembruch U, Reiss I, Gortner L, Weiner CP, Harman CR. Absent umbilical artery end-diastolic velocity in growth-restricted fetuses: a risk factor for neonatal thrombocytopenia. Obstet Gynecol. 2000 Aug;96(2):162-6. doi: 10.1016/s0029-7844(00)00904-2. PMID 10908756
- [Background] Turan OM, Turan S, Gungor S, Berg C, Moyano D, Gembruch U, Nicolaides KH, Harman CR, Baschat AA. Progression of Doppler abnormalities in intrauterine growth restriction. Ultrasound Obstet Gynecol. 2008 Aug;32(2):160-7. doi: 10.1002/uog.5386. PMID 18634130
- [Background] Crimmins S, Desai A, Block-Abraham D, Berg C, Gembruch U, Baschat AA. A comparison of Doppler and biophysical findings between liveborn and stillborn growth-restricted fetuses. Am J Obstet Gynecol. 2014 Dec;211(6):669.e1-10. doi: 10.1016/j.ajog.2014.06.022. Epub 2014 Jun 12. PMID 24931475
- [Background] Caradeux J, Martinez-Portilla RJ, Basuki TR, Kiserud T, Figueras F. Risk of fetal death in growth-restricted fetuses with umbilical and/or ductus venosus absent or reversed end-diastolic velocities before 34 weeks of gestation: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Feb;218(2S):S774-S782.e21. doi: 10.1016/j.ajog.2017.11.566. Epub 2017 Dec 9. PMID 29233550
- [Background] Ferrazzi E, Bozzo M, Rigano S, Bellotti M, Morabito A, Pardi G, Battaglia FC, Galan HL. Temporal sequence of abnormal Doppler changes in the peripheral and central circulatory systems of the severely growth-restricted fetus. Ultrasound Obstet Gynecol. 2002 Feb;19(2):140-6. doi: 10.1046/j.0960-7692.2002.00627.x. PMID 11876805
- [Background] Hecher K, Bilardo CM, Stigter RH, Ville Y, Hackeloer BJ, Kok HJ, Senat MV, Visser GH. Monitoring of fetuses with intrauterine growth restriction: a longitudinal study. Ultrasound Obstet Gynecol. 2001 Dec;18(6):564-70. doi: 10.1046/j.0960-7692.2001.00590.x. PMID 11844190
- [Background] Baschat AA, Gembruch U, Harman CR. The sequence of changes in Doppler and biophysical parameters as severe fetal growth restriction worsens. Ultrasound Obstet Gynecol. 2001 Dec;18(6):571-7. doi: 10.1046/j.0960-7692.2001.00591.x. PMID 11844191
- [Background] Baschat AA, Galan HL, Bhide A, Berg C, Kush ML, Oepkes D, Thilaganathan B, Gembruch U, Harman CR. Doppler and biophysical assessment in growth restricted fetuses: distribution of test results. Ultrasound Obstet Gynecol. 2006 Jan;27(1):41-47. doi: 10.1002/uog.2657. PMID 16323151
- [Background] Lees CC, Marlow N, van Wassenaer-Leemhuis A, Arabin B, Bilardo CM, Brezinka C, Calvert S, Derks JB, Diemert A, Duvekot JJ, Ferrazzi E, Frusca T, Ganzevoort W, Hecher K, Martinelli P, Ostermayer E, Papageorghiou AT, Schlembach D, Schneider KT, Thilaganathan B, Todros T, Valcamonico A, Visser GH, Wolf H; TRUFFLE study group. 2 year neurodevelopmental and intermediate perinatal outcomes in infants with very preterm fetal growth restriction (TRUFFLE): a randomised trial. Lancet. 2015 May 30;385(9983):2162-72. doi: 10.1016/S0140-6736(14)62049-3. Epub 2015 Mar 5. PMID 25747582
- [Background] Sharp A, Cornforth C, Jackson R, Harrold J, Turner MA, Kenny LC, Baker PN, Johnstone ED, Khalil A, von Dadelszen P, Papageorghiou AT, Alfirevic Z; STRIDER group. Maternal sildenafil for severe fetal growth restriction (STRIDER): a multicentre, randomised, placebo-controlled, double-blind trial. Lancet Child Adolesc Health. 2018 Feb;2(2):93-102. doi: 10.1016/S2352-4642(17)30173-6. Epub 2017 Dec 7. PMID 30169244
- [Background] Ylikorkala O, Makila UM, Kaapa P, Viinikka L. Maternal ingestion of acetylsalicylic acid inhibits fetal and neonatal prostacyclin and thromboxane in humans. Am J Obstet Gynecol. 1986 Aug;155(2):345-9. doi: 10.1016/0002-9378(86)90823-9. PMID 3526896
- [Background] Parker CR Jr, Hauth JC, Goldenberg RL, Cooper RL, Dubard MB. Umbilical cord serum levels of thromboxane B2 in term infants of women who participated in a placebo-controlled trial of low-dose aspirin. J Matern Fetal Med. 2000 Jul-Aug;9(4):209-15. doi: 10.1002/1520-6661(200007/08)9:43.0.CO;2-S. PMID 11048830
- [Background] Trudinger BJ, Cook CM, Thompson RS, Giles WB, Connelly A. Low-dose aspirin therapy improves fetal weight in umbilical placental insufficiency. Am J Obstet Gynecol. 1988 Sep;159(3):681-5. doi: 10.1016/s0002-9378(88)80034-6. PMID 3048102
- [Background] Newnham JP, Godfrey M, Walters BJ, Phillips J, Evans SF. Low dose aspirin for the treatment of fetal growth restriction: a randomized controlled trial. Aust N Z J Obstet Gynaecol. 1995 Nov;35(4):370-4. doi: 10.1111/j.1479-828x.1995.tb02144.x. PMID 8717556
- [Background] McCowan LM, Harding J, Roberts A, Barker S, Ford C, Stewart A. Administration of low-dose aspirin to mothers with small for gestational age fetuses and abnormal umbilical Doppler studies to increase birthweight: a randomised double-blind controlled trial. Br J Obstet Gynaecol. 1999 Jul;106(7):647-51. doi: 10.1111/j.1471-0528.1999.tb08362.x. PMID 10428519
- [Background] Ali MK, Abbas AM, Yosef AH, Bahloul M. The effect of low-dose aspirin on fetal weight of idiopathic asymmetrically intrauterine growth restricted fetuses with abnormal umbilical artery Doppler indices: a randomized clinical trial. J Matern Fetal Neonatal Med. 2018 Oct;31(19):2611-2616. doi: 10.1080/14767058.2017.1350160. Epub 2017 Jul 11. PMID 28670938
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Baschat AA, Cosmi E, Bilardo CM, Wolf H, Berg C, Rigano S, Germer U, Moyano D, Turan S, Hartung J, Bhide A, Muller T, Bower S, Nicolaides KH, Thilaganathan B, Gembruch U, Ferrazzi E, Hecher K, Galan HL, Harman CR. Predictors of neonatal outcome in early-onset placental dysfunction. Obstet Gynecol. 2007 Feb;109(2 Pt 1):253-61. doi: 10.1097/01.AOG.0000253215.79121.75. PMID 17267821
- [Background] Sharp A, Jackson R, Cornforth C, Harrold J, Turner MA, Kenny L, Baker PN, Johnstone ED, Khalil A, von Dadelszen P, Papageorghiou AT, Alfirevic Z. A prediction model for short-term neonatal outcomes in severe early-onset fetal growth restriction. Eur J Obstet Gynecol Reprod Biol. 2019 Oct;241:109-118. doi: 10.1016/j.ejogrb.2019.08.007. Epub 2019 Aug 16. PMID 31499415
- [Background] Baschat AA. Neurodevelopment following fetal growth restriction and its relationship with antepartum parameters of placental dysfunction. Ultrasound Obstet Gynecol. 2011 May;37(5):501-14. doi: 10.1002/uog.9008. PMID 21520312
- [Background] Pardey J, Moulden M, Redman CW. A computer system for the numerical analysis of nonstress tests. Am J Obstet Gynecol. 2002 May;186(5):1095-103. doi: 10.1067/mob.2002.122447. PMID 12015543
- [Background] Baschat AA, Kush M, Berg C, Gembruch U, Nicolaides KH, Harman CR, Turan OM. Hematologic profile of neonates with growth restriction is associated with rate and degree of prenatal Doppler deterioration. Ultrasound Obstet Gynecol. 2013 Jan;41(1):66-72. doi: 10.1002/uog.12322. Epub 2012 Dec 14. PMID 23065842